CLINICAL TRIAL: NCT02085200
Title: The Effect of Scapular Stabilization During Horizontal Adduction Stretching on Passive Internal Rotation and Posterior Shoulder Tightness in Young Female Volleyball Athletes.
Brief Title: Scapular Stabilization During Manual Horizontal Adduction Stretches and Its Effect on Increasing Posterior Shoulder Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: Southeastern Orthopedics Sports Medicine and Shoulder Center (Unknown); Triangle Volleyball, Inc. (Industry)
Responsible Party: Principal Investigator, Paul Salamh, Director of Rehabilitation at Southeastern Orthopedics Sports Medicine and Shoulder Center, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 04111311
Record Dates: First submitted 2014-03-07; First posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Posterior Shoulder Tightness
Keywords: glenohumeral internal rotation deficit; overhead athlete; shoulder exercise; posterior glenohumeral capsule; posteroinferior glenohumeral ligament; posterior rotator cuff

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Horizontal adduction stretch without scapular stabilization (Other): Scapular stabilization is not provided during a manual horizontal adduction stretch of the shoulder. Each stretch is held for 25 seconds and repeated for a total of 3 times.
  Interventions: Other: Horizontal adduction stretch without scapular stabilization
- Horizontal adduction with scapular stabilization (Other): Scapular stabilization is provided during a manual horizontal adduction stretch of the shoulder. Each stretch is held for 25 seconds and repeated for a total of 3 times.
  Interventions: Other: horizontal adduction stretch with scapular stabilization

INTERVENTIONS:
Other: horizontal adduction stretch with scapular stabilization — Scapular is stabilized during manual horizontal adduction stretch
  Arms: Horizontal adduction with scapular stabilization
Other: Horizontal adduction stretch without scapular stabilization — Scapula stabilization is not performed during horizontal adduction stretch
  Arms: Horizontal adduction stretch without scapular stabilization

SUMMARY:
The purpose of this study is to determine if stabilizing the scapula (shoulder blade) during a common shoulder stretch is more effective at improving shoulder range of motion than not stabilizing the scapula. Investigators hypothesize that scapular stabilization during horizontal adduction stretching will demonstrate greater gains in shoulder range of motion than stretching without scapular stabilization.

ELIGIBILITY:
Inclusion Criteria:

* athletes with at least two years of volleyball experience
* athletes with no current shoulder pain
* athletes between the ages of 15 and 21
* athletes with a 10 degree or greater difference in internal rotation between shoulders

Exclusion Criteria:

* athletes currently experiencing shoulder pain
* athletes having less than two years of volleyball experience
* athletes not meting inclusion criteria

Ages: 15 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in Posterior Shoulder Tightness | Change from baseline posterior shoulder tightness to immediately following manual stretching. The baseline is measured, followed by 3 stretches held for 25 seconds and then the follow up measure is taken. This is the conclusion of this measure.
  An inclinometer is used to measure posterior shoulder tightness.

SECONDARY OUTCOMES:
Change in Internal Rotation | Change from baseline internal rotation to immediately following manual stretching. The baseline is measured, followed by 3 stretches held for 25 seconds and then the follow up measure is taken. This is the conclusion of this measure.
  An inclinometer is used to measure internal rotation

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Salamh, PT,DPT,PhD(c), Principal Investigator — Nova Southeastern University and Southeastern Orthopedics Sports Medicine and Shoulder Center
Locations (1):
- Triangle Volleyball Club Inc., Morrisville, North Carolina, United States

REFERENCES:
- [Derived] Salamh PA, Kolber MJ, Hanney WJ. Effect of scapular stabilization during horizontal adduction stretching on passive internal rotation and posterior shoulder tightness in young women volleyball athletes: a randomized controlled trial. Arch Phys Med Rehabil. 2015 Feb;96(2):349-56. doi: 10.1016/j.apmr.2014.09.038. Epub 2014 Oct 23. PMID 25450120